CLINICAL TRIAL: NCT07388511
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Elenestinib on the Pharmacokinetics of Midazolam and Combined Oral Contraceptives, Levonorgestrel/Ethinyl Estradiol, in Healthy Adult Female Participants
Brief Title: A Study of Elenestinib in Healthy Adult Female Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BLU-263-0104
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Midazolam; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elenestinib, Midazolam, and Levonorgestrel/Ethinyl Estradiol (Experimental)
  Interventions: Drug: Elenestinib; Drug: Midazolam; Drug: Levonorgestrel/Ethinyl Estradiol

INTERVENTIONS:
Drug: Elenestinib — Specified dose on specified days
Drug: Midazolam — Specified dose on specified days
Drug: Levonorgestrel/Ethinyl Estradiol — Specified dose on specified days

SUMMARY:
The main objectives of this study are to determine the effect of elenestinib on the pharmacokinetic parameters (how the drug is absorbed, distributed, and processed by the body) of midazolam, and to determine the effect of elenestinib on the pharmacokinetic parameters of levonorgestrel/ethinyl estradiol, when given as a combined oral contraceptive.

Healthy adult participants will receive midazolam and levonorgestrel/ethinyl estradiol with and without elenestinib and have blood samples taken.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, adult, female, 18-65 years of age, inclusive, at the screening visit that meet either of the following criteria:
* Postmenopausal female, defined as amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status at the screening visit (note that participants may have had hysterectomy, bilateral salpingectomy, or bilateral tubal ligation).
* Female status-post bilateral oophorectomy.
* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 6 months prior to the first dosing.
* BMI ≥ 18.0 and ≤ 35.0 kg/m2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and electrocardiograms (ECGs), as deemed by the principal investigator (PI) or designee.

Key Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History or presence of alcohol or drug abuse (except for the occasional use of cannabis products) within the past 1 years prior to the first dosing.
* History or presence of cannabis use within the past 3 months prior to the first dosing.
* History or presence of hypersensitivity or idiosyncratic reaction to elenestinib, midazolam, combined oral contraceptive (levonorgestrel/ethinyl estradiol), or related compounds.
* Unable to refrain from or anticipates the use of:
* Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing.
* Any drugs known to be moderate or strong inducers of CYP3A4 enzymes and/or P-gp beginning at least 28 days prior to first dosing.
* Any drugs known to increase or decrease levels of SHBG, including any oral, topical, or intravaginal hormone-containing product, within 12 weeks prior to the first dosing.

Other protocol-defined inclusion and exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (AUC0-t) | Up to 27 days
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) | Up to 27 days
Percent of AUC0-inf extrapolated (AUC%extrap) | Up to 27 days
Maximum observed concentration (Cmax) | Up to 27 days
Time to reach Cmax (Tmax) | Up to 27 days
Apparent first-order terminal elimination half-life (t1/2) | Up to 27 days
Apparent total plasma clearance after oral administration (CL/F) | Up to 27 days
Apparent volume of distribution during the terminal elimination phase after oral administration (Vz/F) | Up to 27 days

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From first dose to date of last dose plus 30 days (up to approximately 7 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States